CLINICAL TRIAL: NCT03216174
Title: Pilot Study of Non-exposure Simple Suturing EFTR (NESS-EFTR) With Sentinel Lymph Node Navigation for Early Gastric Cancer (Senorita3-pilot)
Brief Title: Pilot Study of Non-exposure Simple Suturing EFTR With Sentinel Lymph Node Navigation for EGC (Senorita3-pilot)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Chan Gyoo Kim, Senior scientist, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2017-0088
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NESS-EFTR (Experimental): This arm will be received non-exposure simple suturing endoscopic full-thickness resection after sentinel lymph node navigation
  Interventions: Procedure: NESS-EFTR

INTERVENTIONS:
Procedure: NESS-EFTR — NESS-EFTR includes steps of laparoscopic seromuscular suturing, EFTR of the inverted stomach wall, and endoscopic mucosal suturing with endoloops and clips.

SUMMARY:
Laparoscopic sentinel lymph node dissection and stomach preserving surgery in early gastric cancer is less invasive method which can increase quality of life. Current stomach preserving surgery after sentinel lymph node dissection produce transmural communication and expose the tumor to the peritoneum during operation. An endoscopic full-thickness resection method with a simple suturing technique that does not expose the gastric mucosa to the peritoneum (non-exposure simple suturing, NESS) was recently developed.

This is the pilot study to prove the feasibility of NESS-EFTR with sentinel node navigation in early gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* single lesion of adenocarcinoma in preoperative endoscopic biopsy
* clinical stage T1N0 in the preoperative evaluation of endoscopy and computed tomography
* tumor size: less than 3cm in differentiated type, less than 2cm in undifferentiated type
* location: 2cm far from the pylorus or cardia
* aged 20 to 80
* ECOG 0 or 1
* patient who signed the agreement
* patient who is suspected to underwent laparoscopy assisted gastrectomy

Exclusion Criteria:

* indication of endoscopic submucosal resection
* inoperable due to poor cardiac, pulmonary function
* pregnant
* having allergic reaction, previous upper abdominal surgery except laparoscopic cholecystectomy, previous radiation therapy to upper abdomen
* diagnosed as malignancy within 5 years except carcinoma in situ of cervix cancer and thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-11 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete resection | 3 months
  single piece resection with clear resection margin

CONTACTS AND LOCATIONS:
Overall Officials: Chan Gyoo Kim, M.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eom BW, Kim CG, Kook MC, Yoon HM, Ryu KW, Kim YW, Rho JY, Kim YI, Lee JY, Choi IJ. Non-exposure Simple Suturing Endoscopic Full-thickness Resection with Sentinel Basin Dissection in Patients with Early Gastric Cancer: the SENORITA 3 Pilot Study. J Gastric Cancer. 2020 Sep;20(3):245-255. doi: 10.5230/jgc.2020.20.e22. Epub 2020 Jul 6. PMID 33024581